CLINICAL TRIAL: NCT03037333
Title: Prospective Analysis in the EMERGEncy Between TransVenous Cardiac PACIng Guided by Fluoroscopy Versus Echocardiogram
Brief Title: Analysis in the EMERGEncy Between TransVenous Cardiac PACIng Guided by Fluoroscopy Versus Echocardiogram
Acronym: EMERG-TV-PAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSInCor-EMERG-TV-PAC
Record Dates: First submitted 2017-01-18; First posted 2017-01-31 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Bradycardia
Keywords: echocardiogram; Electrocardiogram: Electrical Alternans; fluoroscopy
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluoroscopy (Other)
  Interventions: Procedure: Transvenous cardiac pacing guided by fluoroscopy
- ECG/ECHO (Other)
  Interventions: Procedure: Transvenous cardiac pacing guided by ECG/ECHO

INTERVENTIONS:
Procedure: Transvenous cardiac pacing guided by fluoroscopy — Transvenous cardiac estimulation
  Arms: fluoroscopy
Procedure: Transvenous cardiac pacing guided by ECG/ECHO — Transvenous cardiac estimulation
  Arms: ECG/ECHO

SUMMARY:
A lot of questions about use of temporary transvenous pacing still remain obscure and there is no effective comparison between use of fluoroscopy versus electrocardiogram/echocardiogram in patients with bradicardias. The aim of the study is to evaluate how long does it take to start the correct cardiac stimulation with transvenous pacing in patients with bradicardias comparing use of fluoroscopy versus electrocardiogram/echocardiogram and compare rates of complications between two methods.

DETAILED DESCRIPTION:
Approximately 150 subjects will be recruited over a planned recruitment period of 18 months. Patients will be submitted to ecchocardiogram using Philips Envisor, and electrocardiogram with Philips Healthcare PageWriter TC30.

ELIGIBILITY:
Inclusion Criteria:

* adult males and females aged > 18 years
* symptomatic bradicardia
* informed consent signed.

Exclusion Criteria:

* pregnancy
* hemodynamic instability (pulmonary congestion / systolic arterial pressure lower than 90 mmHg)
* body mass index greater than 40 kg/ m2
* use of oral anticoagulation
* acute coronary syndromes
* left ventricle ejection fraction < 45%
* presence of any kind of cardiac stimulation device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 1 week
infection | 1 week
  Incidence of infection assessed by a clinical diagnosis
hematoma > 5 cm | 1 week
  image
cardiac perforation | 1 week
  Incidence of cardiac perforation assessed by a clinical diagnosis
pneumothorax | 1 week
  Incidence of pneumothorax assessed by a clinical diagnosis
ventricular tachycardia | 1 week
  Incidence of ventricular tachycardia assessed by an ECG test
loss of capture | 1 week
  Incidence of loss of capture assessed by an ECG test
venous thrombosis | 1 week
  Incidence of venous thrombosis assessed by an ultrasound
any complication the delays definitive pacemaker > 48 hours | 1 week
  clinical diagnosis

SECONDARY OUTCOMES:
Time to start the correct cardiac stimulation with transvenous pacing | 1 week
  minutes scale
rates of success | 1 week
  ECG test

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Soeiro, MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Esmaiel A, Hassan J, Blenkhorn F, Mardigyan V. The Use of Ultrasound to Improve Axillary Vein Access and Minimize Complications during Pacemaker Implantation. Pacing Clin Electrophysiol. 2016 May;39(5):478-82. doi: 10.1111/pace.12833. Epub 2016 Mar 23. PMID 26880272
- [Result] Reusz G, Csomos A. The role of ultrasound guidance for vascular access. Curr Opin Anaesthesiol. 2015 Dec;28(6):710-6. doi: 10.1097/ACO.0000000000000245. PMID 26539789
- [Result] Bouaziz H, Zetlaoui PJ, Pierre S, Desruennes E, Fritsch N, Jochum D, Lapostolle F, Pirotte T, Villiers S. Guidelines on the use of ultrasound guidance for vascular access. Anaesth Crit Care Pain Med. 2015 Feb;34(1):65-9. doi: 10.1016/j.accpm.2015.01.004. Epub 2015 Mar 5. PMID 25829319
- See also: Related Info — http://journals.sagepub.com/doi/pdf/10.1177/2048872615572598
- See also: Related Info — http://onlinelibrary.wiley.com/doi/10.1111/jce.12005/abstract
- See also: Related Info — https://cardiovascularultrasound.biomedcentral.com/articles/10.1186/s12947-015-0004-9